CLINICAL TRIAL: NCT03888651
Title: An Investigation of Postoperative Chronic Opioid Use and Its Associations With Other Clinical Factors Among Patients With Head and Neck Cancers
Brief Title: Clinical Data Collection in Studying Clinical Factors Associated With Post-Surgery Chronic Opioid Use in Patients With Head and Neck Cancers
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2018-0740; NCI-2018-03357 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0740 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2019-01-16; First posted 2019-03-25 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaires, quality of life assessment): Patients complete questionnaires and quality of life assessments over 10-15 minutes at pre-surgery, after-surgery, at discharge, within 2-3 weeks after surgery, and within 90 days after surgery.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Complete quality of life assessment
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This trial studies the risk of developing disorders associated with chronic opioid use post-surgery in patients with head and neck cancers. Clinical data collection may help doctors to learn how often and how likely disorders associated with the use of opioid pain medication may occur in patients with head and neck cancer who are having surgery as part of their treatment plan.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess prevalence of chronic opioid use and severity of symptom burden (M. D. Anderson Symptom Inventory-Head and Neck [MDASI-HN]) in patients undergoing surgery of head/neck cancer.

SECONDARY OBJECTIVES:

I. To investigate the extent of association of chronic opioid use with risk of opioid use disorder (as assessed by Screener and Opioid Assessment for Patients with Pain[SOAPP-14] and Cut down, Annoyed, Guilty and Eye Opener [CAGE] scores) and psychosocial factors (as assessed by MDASI).

II. To assess frequency of positive risk of opioid use disorder as assessed by Screener and Opioid Assessment for Patients tool (SOAPP-14) and CAGE-adapted to include drugs (AID).

III. Assess frequency of aberrant opioid use behaviors. IV. Assess frequency of post-operative complications.

OUTLINE:

Patients complete questionnaires and quality of life assessments over 10-15 minutes at pre-surgery, after-surgery, at discharge, within 2-3 weeks after surgery, and within 90 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with head and neck cancer scheduled for combined head and neck surgery - plastic surgery free flap
* Competent to give informed consent
* Ability to read and write in English

Exclusion Criteria:

* Patient not willing to participate
* Not competent to give informed consent
* Inability to read and write in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Participants
Sampling Method: Non-Probability Sample
Enrollment: 125 (Estimated)
Dates: Start 2019-01-25 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Rate of chronic opioid use | At 90 days after surgery
  Rate of chronic opioid use will be measured by the association of chronic opioid use with that of the risk of opioid misuse Screener and Opioid Assessment for Patients tool (SOAPP-14)
Severity of symptom burden | At 90 days after surgery
  Will be measured by MDASI.
Association of chronic opioid use | At 90 days after surgery
  Association of chronic opioid use with that of the CAGE-AID scores

SECONDARY OUTCOMES:
Risk of opioid use assessed | Up to 90 days after surgery
  Screener and Opioid Assessment for Patients with Pain[SOAPP-14] Score of greater than or equal 7 is considered as risk factor for opioid misuse.
Frequency of positive risk of opioid use disorder | Up to 90 days post surgery
  Will be assessed by Screener and Opioid Assessment for Patients with Pain[SOAPP-14.
Frequency of aberrant opioid use behaviors | Up to 90 days post surgery
  Correlation between categorical variables will be evaluated using Chisquare test or Fisher's exact test.
Frequency of post-operative complications | Up to 90 days post surgery
  Correlation between categorical variables will be evaluated using Chisquare test or Fisher's exact test
Risk of opioid use will be assessed by CAGE-AID | Up to 90 days post surgery
  CAGE-AID: Score of greater than or equal 2 is considered as risk factor for opioid misuse
Frequency of positive risk of opioid use disorder | Up to 90 days post surgery
  Will be assessed by CAGE-adapted to include drugs (AID).

CONTACTS AND LOCATIONS:
Overall Officials: Lakshmi Koyyalagunta, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org